CLINICAL TRIAL: NCT03061292
Title: A Randomized, Controlled Trial on Patients Undergoing Cardiac Implantable Electronic Device Implantation With Local Anaesthesia and Sedation With and Without Pectoral Nerve Block
Brief Title: Cardiac Implantable Electronic Device Implantation With and Without Pectoral Nerve Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Other
Other Study IDs: PECS
Record Dates: First submitted 2017-02-14; First posted 2017-02-23 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Cardiac IED Implantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pectoral Nerve Block (Experimental): Patients undergoing cardiac implantable electronic device implantation with local anaesthesia and sedation with pectoral nerve block
  Interventions: Procedure: Pectoral Nerve Block
- Without Pectoral Nerve Block (Sham Comparator): Patients undergoing cardiac implantable electronic device implantation with local anaesthesia and sedation without pectoral nerve block
  Interventions: Procedure: Without Pectoral Nerve Block

INTERVENTIONS:
Procedure: Pectoral Nerve Block
  Arms: Pectoral Nerve Block
Procedure: Without Pectoral Nerve Block
  Arms: Without Pectoral Nerve Block

SUMMARY:
Implantation of cardiac implantable electronic devices are generally carried out using intermittent intravenous conscious sedation combined with local anaesthesia. The main advantage of this technique is in avoiding the potential risks of general anaesthesia. However, the use of this Sedation - Local Anaesthesia technique is not without complications. Peri -procedural hypoxaemia and hypotension are well recognised complications of this technique.

The pectoral nerves (Pecs) blocks are novel techniques to block the pectoral, intercostobrachial, third to sixth intercostals, and the long thoracic nerves. PECS block targets the lateral and median pectoral nerves at an interfascial plane between the pectoralis major and minor muscles.

A case report by Fujiwara et al has described the use of this technique to provide good analgesia during and after these implantation procedures surgery. Pectoral nerves block along with minimal sedation has been used as a safe technique in our local set up as well.

Hence, we propose a randomized, single center, controlled trial on patients undergoing cardiac implantable electronic device implantation with local anaesthesia and sedation with and without Pectoral Nerve Block.

DETAILED DESCRIPTION:
Intervention group:

Pectoral nerve block will be performed by anaesthetist (not blinded) in cardiac catheterization laboratory using ultrasound guidance and strict aseptic technique.

Control group:

A sham "block" will be performed by anaesthetist in cardiac catheterization laboratory using strict aseptic technique.

Patients of both groups will be monitored by the Cardiologist ( performing the procedure) and the Nurse from the monitoring room.

A minimum period of 15 minutes will be allowed following the block, prior to device implantation procedure by cardiologist.

Numeric rating scale (NRS) will be used for assessment of pain. The assessment will be carried out at every 15 minutes from the start of the procedure till the end of the procedure (0, 15, 30, 45, 60 minutes etc) and also at specific time points. Numerical rating scale will also be assessed when the patient experiences pain at any point and in the recovery room (0, 15, 30 and if needed, 45, 60 minutes).

Further post-operative pain scores will be collected at 4 hours and 8 hours post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilled the indication for CIED implantation as defined in 2008 guidelines for device-based therapy of cardiac rhythm abnormalities

Exclusion Criteria:

* Pregnant
* Those who receives subcutaneous implantable cardioverter defibrillator
* Vulnerable subjects (children, prisoners, cognitive impaired persons)
* Known history of allergy to local anaesthetic medications

Ages: 21 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-07-25 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Total dose of sedation used | 2 years
Incidence of hypoxia, hypotension and hypopnea in the perioperative period | 2 years
Perioperative sedation scores | 2 years
Perioperative pain scores | 2 years
Post-anaesthetic discharge score | 2 years

SECONDARY OUTCOMES:
Procedurist satisfaction scores | 2 years
Patient satisfaction scores | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided